CLINICAL TRIAL: NCT03481660
Title: A Two-Year, Two-Arm, Randomized, Double Masked, Multicenter, Phase III Study Assessing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Adult Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: A Study of the Efficacy and Safety of Brolucizumab vs. Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: KITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRTH258B2302; 2017-003960-11 (EudraCT Number)
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; intravitreal injection; brolucizumab; aflibercept; double-masked
MeSH Terms: interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): Brolucizumab 6 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule
  Interventions: Drug: Brolucizumab
- Aflibercept 2 mg (Active Comparator): Aflibercept 2 mg/0.05 mL, as labeled, 5 loading doses, with subsequent doses every 8 weeks
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — Intravitreal injection
  Other Names: RTH258, ESBA1008
  Arms: Brolucizumab 6 mg
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
This was a Phase III, randomized, double-masked, multi-center, active-controlled, two-arm study designed to evaluate the efficacy and safety of brolucizumab 6 mg compared to the active control, aflibercept 2 mg used per authorized label, in subjects with visual impairment due to diabetic macular edema (DME).

DETAILED DESCRIPTION:
The study included a screening period of up to 2 weeks to assess eligibility, followed by a double-masked treatment period (Day 1 to Week 96). The baseline visit was defined as Day 1/Visit 1, and end of treatment visit as Visit 27 (Week 96). After the last treatment visit, there was a post-treatment follow-up period from Week 96 to Week 100 and an exit visit at Week 100. Subjects were assigned to one of two treatment arms in a 1:1 ratio: brolucizumab 6 mg/0.05 mL (5 loading doses each administered every 6 weeks (q6w) during loading phase then q12w/q8w during maintenance phase with an option to extend treatment interval by 4 weeks during the second year) or aflibercept 2 mg/0.05 mL (5 loading doses each administered every 4 weeks (q4w) during loading phase then q8w during maintenance phase).

Disease activity assessments (DAAs) were conducted by the masked investigator for both treatment arms at Week 32 and Week 36, i.e., 8 and 12 weeks after the end of the loading phase for subjects receiving brolucizumab, and at Week 48, Week 60 and Week 72 (i.e., every 12 weeks). In the brolucizumab arm, subjects who qualified for q12w during this initial q12w interval continued on a q12w treatment frequency unless disease activity was identified at any of the subsequent DAA visits, in which case subjects were switched to a q8w treatment interval until Week 72.

A one-time disease stability assessment was performed by the masked investigator at Week 72 in both treatment arms with the purpose of evaluating the potential for treatment interval extension by 4 weeks. The subjects in the brolucizumab arm who demonstrated disease stability in the one-time assessment at Week 72 under their current assigned treatment regimen (q12w or q8w) were considered for treatment interval extension. To evaluate the adequacy of the individualized q8w, q12w or q16w treatment intervals in the brolucizumab arm, DAAs were performed at every visit from Week 72 up to and including Week 96 (i.e., every 4 weeks) and subjects had their treatment interval modified accordingly. If after Week 72 disease activity had been identified by the masked investigator at a scheduled treatment visit (according to the subject specific treatment schedule q12w or q16w) the subject was assigned to q8w treatment schedule.

ELIGIBILITY:
Key Inclusion Criteria:

General

* Patients must give written informed consent before any study related assessments are performed
* Patients with type 1 or type 2 diabetes mellitus and HbA1c of =< 10% at screening
* Medication for the management of diabetes must have been stable within 3 months prior to randomization and is expected to remain stable during the course of the study

Study Eye

* Visual impairment due to DME with:

  1. BCVA score between 78 and 23 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/320), at screening and baseline
  2. DME involving the center of the macula, with central subfield retinal thickness (measured from RPE to ILM inclusively) of >= 320 micrometers (μm) on SD-OCT at screening If both eyes are eligible, the eye with the worse visual acuity will be selected for study eye. However, the investigator may select the eye with better visual acuity, based on medical reasons or local ethical requirements.

     Key Exclusion Criteria:
* Previous treatment with any anti-VEGF drugs or investigational drugs in the study eye
* Active proliferative diabetic retinopathy in the study eye as per the investigator
* Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the first 12-month study period (e.g., cataract, vitreous hemorrhage, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause)
* Any active intraocular or periocular infection or active intraocular inflammation (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye at screening or baseline
* Structural damage of the fovea in the study eye at screening likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), epiretinal membrane involving fovea or organized hard exudate plaques
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 millimeters mercury (mmHg) on medication or according to investigator's judgment, at screening or baseline
* Neovascularization of the iris in the study eye at screening or baseline
* Evidence of vitreomacular traction in the study eye at screening or baseline which, in the opinion of the investigator, affect visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (68):
- Novartis Investigative Site, Alken, Belgium
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Roskilde
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (11):
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- India (5):
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Riga, Latvia
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Malaysia (2):
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Shah Alam, Selangor
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Gdansk, Poland
- Russia (4):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (4):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Trenčín
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Örebro, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 79 centers in 23 countries: Belgium (1), Bulgaria (3), Czech Republic (3), Denmark (2), Estonia (2), France (12), Germany (7), Hungary (5), India (5), Republic of Korea (6), Latvia (1), Lebanon (3), Lithuania (2), Malaysia (2), Norway (1), Poland (1), Russia (5), Singapore (2), Slovakia (5), Sweden (1), Switzerland (2), Taiwan (3), Turkey (5).
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started (All randomized treated patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF)) | 179 | 181
Completed | 143 | 156
Not Completed | 36 | 25
Not completed — Adverse Event | 5 | 4
Not completed — Death | 13 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 179 | 181 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (10.55) | 62.2 (9.48) | 62.2 (10.01)
Age, Customized [Number; unit: Participants]
  < 65 years | 100 | 102 | 202
  >= 65 years | 79 | 79 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 125
  Male | 120 | 115 | 235
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 163 | 170 | 333
  Unknown or Not Reported | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 48 | 91
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 133 | 132 | 265
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) at Week 52 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The overall BCVA score (number of letters read correctly by the patient) was calculated using the BCVA worksheet 0-100 letter score, with higher score indicating improvement in acuity. A positive change from baseline is a favorable outcome. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale | 10.6 [9.3 to 11.9] | 9.4 [8.1 to 10.7]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA at Week 52; Test type: Non-Inferiority — (4-letter margin) (1-sided); p < 0.001, ANOVA; LS mean difference = 1.2, 95% CI 2-sided [-0.6 to 3.1], Standard Error of Mean 0.94

2. Secondary Outcome: Average Mean Change From Baseline in BCVA Over the Period Week 40 Through Week 52 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The overall BCVA score (number of letters read correctly by the patient) was calculated using the BCVA worksheet 0-100 letter score, with higher score indicating improvement in acuity. A positive change from baseline is a favorable outcome. For each participants, this endpoint was defined as the mean change from baseline to the average value over the period Week 40 through Week 52. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, period Week 40 through Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale | 10.3 [9.1 to 11.5] | 9.4 [8.2 to 10.6]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 40 through Week 52; Test type: Non-Inferiority — (4-letter margin) (1-sided); p < 0.001, ANOVA; LS mean difference = 0.9, 95% CI 2-sided [-0.9 to 2.6], Standard Error of Mean 0.88
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 40 through Week 52; Test type: Superiority; p = 0.164, ANOVA

3. Secondary Outcome: (Brolucizumab Treatment Arm Only): Percentage of Participants Maintained at q12w up to Week 52 and up to q12w/q16w up to Week 100.
Description: The number of participants maintaining every 12 weeks (q12w) treatment status in the Brolucizumab arm was derived based on Kaplan-Meier estimates time-to-first q8w treatment need. Positive treatment status was defined as intravitreal treatment (IVT) injections per planned dosing regimen [every 12 weeks (q12w)].
Time Frame: Week 52, Week 100
Population: Full Analysis Set - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
Percentage of participants
  Week 48 | 50.3 [42.5 to 57.7] |
  Week 96 | 36.8 [29.1 to 45.5] |

4. Secondary Outcome: (Brolucizumab Treatment Arm Only): Percentage of Participants Maintained at q12w up to Week 52 Within Those Patients That Qualified for q12w at Week 36
Description: as for outcome 3
Time Frame: Week 36, Week 52
Population: Full Analysis Set - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 87 | 0
Percentage of participants | 95.1 [87.4 to 98.1] |

5. Secondary Outcome: (Brolucizumab Treatment Arm Only): Percentage of Participants Maintained at q12w/q16w up to Week 100, Within Those Patients That Qualified for q12w at Week 36
Description: Disease activity assessments (DAAs) were performed to identify q8w-need at pre-specified visits (Weeks 32, 36, 48, 60, 72 and every visit from Week 72 through Week 96). Weeks 32 and 36 were the two DAA visits of the initial q12w cycle after the loading phase of the brolucizumab arm. At Week 72 or Week 76 (if DAA/disease stability assessment was missed at Week 72), participants in the brolucizumab were evaluated for an additional 4-week dose regimen extension.
  The number of participants maintaining every 12 weeks (q12w) treatment status in the Brolucizumab arm was derived based on Kaplan-Meier estimates time-to-first q8w treatment need. Positive treatment status was defined as intravitreal treatment (IVT) injections per planned dosing regimen [every 12 weeks (q12w)].
Time Frame: Week 36, Week 100
Population: Full Analysis Set - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 87 | 0
Percentage of participants | 69.6 [57.4 to 78.9] |

6. Secondary Outcome: (Brolucizumab Treatment Arm Only): Percentage of Participants Maintained on q16w up to Week 100 Within the Patients on q12w at Week 68 and on q16w at Week 76
Description: as for outcome 5
Time Frame: Week 68, Week 76, Week 100
Population: Full Analysis Set - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 44 | 0
Percentage of participants | 87.9 [73.3 to 94.8] |

7. Secondary Outcome: (Brolucizumab Treatment Arm Only): Percentage of Participants Re-assigned and Maintained on q12w up to Week 100 Within the Patients on q8w at Week 68 and on q12w at Week 80
Description: as for outcome 5
Time Frame: Week 68, Week 80, Week 100
Population: Full Analysis Set - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 34 | 0
Percentage of participants | 73.1 [54.5 to 85.0] |

8. Secondary Outcome: (Brolucizumab Treatment Arm Only): Number of Participants With Injections Per Planned Dosing Regimen (Every 8, 12 or 16 Weeks)
Description: Reported categorically for the subjects who completed the study treatment period: every 8 weeks (q8w), Every 12 weeks (q12w), Every 16 weeks (q16w)
Time Frame: Week 100
Population: Full Analysis Set. Only participants who completed the study treatment period were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 141 | 0
Participants
  q8w | 74 |
  q12w | 32 |
  q16w | 35 |

9. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Each Visit up to Week 100 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, Week 4, Week 6, Week 8, Week 12, Week 16, Week 18, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56, Week 60, Week 64, Week 68, Week 72, Week 76, Week 80, Week 84, Week 88, Week 92, Week 96, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale
  Week 4 | 5.1 [4.3 to 6.0] | 4.2 [3.4 to 5.1]
  Week 6 | 6.8 [5.9 to 7.6] | 5.9 [5.0 to 6.7]
  Week 8 | 7.8 [6.9 to 8.7] | 6.7 [5.8 to 7.5]
  Week 12 | 8.6 [7.6 to 9.5] | 7.7 [6.7 to 8.6]
  Week 16 | 9.0 [7.9 to 10.1] | 8.3 [7.2 to 9.5]
  Week 18 | 9.2 [8.0 to 10.3] | 9.2 [8.0 to 10.3]
  Week 20 | 9.6 [8.4 to 10.8] | 9.4 [8.2 to 10.6]
  Week 24 | 10.0 [8.8 to 11.2] | 8.7 [7.5 to 9.9]
  Week 28 | 9.8 [8.6 to 11.1] | 9.4 [8.2 to 10.6]
  Week 32 | 10.3 [9.1 to 11.5] | 8.9 [7.7 to 10.1]
  Week 36 | 9.6 [8.4 to 10.9] | 9.4 [8.2 to 10.7]
  Week 40 | 9.9 [8.7 to 11.2] | 9.2 [7.9 to 10.4]
  Week 44 | 10.6 [9.3 to 11.8] | 9.5 [8.3 to 10.8]
  Week 48 | 10.1 [8.8 to 11.3] | 9.6 [8.3 to 10.9]
  Week 52 | 10.6 [9.3 to 11.9] | 9.4 [8.1 to 10.7]
  Week 56 | 10.7 [9.3 to 12.0] | 9.5 [8.2 to 10.9]
  Week 60 | 10.5 [9.1 to 11.9] | 9.3 [8.0 to 10.7]
  Week 64 | 11.0 [9.7 to 12.3] | 9.5 [8.2 to 10.8]
  Week 68 | 11.0 [9.6 to 12.3] | 9.5 [8.2 to 10.8]
  Week 72 | 11.0 [9.6 to 12.3] | 9.4 [8.1 to 10.8]
  Week 76 | 10.5 [9.2 to 11.8] | 9.8 [8.4 to 11.1]
  Week 80 | 10.2 [8.9 to 11.6] | 9.4 [8.1 to 10.8]
  Week 84 | 10.9 [9.4 to 12.4] | 8.9 [7.4 to 10.4]
  Week 88 | 10.7 [9.1 to 12.4] | 8.6 [7.0 to 10.2]
  Week 92 | 10.7 [9.1 to 12.2] | 9.3 [7.7 to 10.8]
  Week 96 | 10.7 [9.1 to 12.3] | 8.5 [6.8 to 10.1]
  Week 100 | 10.9 [9.3 to 12.6] | 8.4 [6.7 to 10.1]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA at Week 52; Test type: Other — Treatment Difference; LS mean difference = 1.2, 95% CI 2-sided [-0.6 to 3.1], Standard Error of Mean 0.94
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA at Week 100; Test type: Other — Treatment Difference; LS mean difference = 2.6, 95% CI 2-sided [0.2 to 4.9], Standard Error of Mean 1.21

10. Secondary Outcome: Average Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Over the Period Week 4 to Week 52/100 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The overall BCVA score (number of letters read correctly by the patient) was calculated using the BCVA worksheet 0-100 letter score, with higher score indicating improvement in acuity. A positive change from baseline is a favorable outcome. For each participants, this endpoint was defined as the mean change from baseline to the average value over the periods: Week 4 through Week 52, Week 4 through Week 100. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, period Week 4 through Week 52, period Week 4 through Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale
  period Week 4 through Week 52 | 9.1 [8.2 to 10.1] | 8.4 [7.4 to 9.3]
  period Week 4 through Week 100 | 9.8 [8.8 to 10.9] | 8.7 [7.7 to 9.8]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 4 through Week 52; Test type: Other — Treatment difference; LS mean difference = 0.8, 95% CI 2-sided [-0.6 to 2.1], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 4 through Week 100; Test type: Other — Treatment difference; LS mean difference = 1.1, 95% CI 2-sided [-0.4 to 2.6], Standard Error of Mean 0.78

11. Secondary Outcome: Average Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Over the Period Week 20 to Week 52/100 and Week 28 to Week 52/100 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The overall BCVA score (number of letters read correctly by the patient) was calculated using the BCVA worksheet 0-100 letter score, with higher score indicating improvement in acuity. A positive change from baseline is a favorable outcome. For each participants, this endpoint was defined as the mean change from baseline to the average value over the periods: Week 20 through Week 52, Week 20 through Week 100, Week 28 through Week 52, Week 28 through Week 100. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, period Week 20 through Week 52, period Week 20 through Week 100, period Week 28 through Week 52, period Week 28 through Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale
  period Week 20 through Week 52 | 10.1 [8.9 to 11.2] | 9.3 [8.1 to 10.4]
  period Week 20 through Week 100 | 10.4 [9.2 to 11.7] | 9.2 [8.0 to 10.4]
  period Week 28 through Week 52 | 10.1 [9.0 to 11.3] | 9.4 [8.2 to 10.5]
  period Week 28 through Week 100 | 10.5 [9.3 to 11.7] | 9.2 [8.0 to 10.5]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 20 through Week 52; Test type: Other — Treatment difference; LS mean difference = 0.8, 95% CI 2-sided [-0.9 to 2.4], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 28 through Week 52; Test type: Other — Treatment difference; LS mean difference = 0.8, 95% CI 2-sided [-0.9 to 2.5], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 20 through Week 100; Test type: Other — Treatment difference; LS mean difference = 1.2, 95% CI 2-sided [-0.5 to 2.9], Standard Error of Mean 0.87
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 28 through Week 100; Test type: Other — Treatment difference; LS mean difference = 1.3, 95% CI 2-sided [-0.5 to 3.0], Standard Error of Mean 0.89

12. Secondary Outcome: Average Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Over the Period Week 88 to 100 for the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The overall BCVA score (number of letters read correctly by the patient) was calculated using the BCVA worksheet 0-100 letter score, with higher score indicating improvement in acuity. A positive change from baseline is a favorable outcome. For each participants, this endpoint was defined as the mean change from baseline to the average value over the period Week 88 through Week 100. BCVA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, period Week 88 through Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Scores on a scale | 10.8 [9.2 to 12.3] | 8.7 [7.1 to 10.2]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; BCVA over period Week 88 through Week 100; Test type: Other — Treatment difference; LS mean difference = 2.1, 95% CI 2-sided [-0.1 to 4.3], Standard Error of Mean 1.12

13. Secondary Outcome: Percentage of Participants Who Gained >= 5 Letters in BCVA From Baseline or Reached BCVA >= 84 Letters at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 49.2 [41.6 to 56.7] | 46.4 [39.0 to 54.0]
  Week 6 | 62.0 [54.5 to 69.1] | 62.4 [54.9 to 69.5]
  Week 8 | 67.6 [60.2 to 74.4] | 63.5 [56.1 to 70.5]
  Week 12 | 70.9 [63.7 to 77.5] | 73.5 [66.4 to 79.8]
  Week 16 | 71.5 [64.3 to 78.0] | 73.5 [66.4 to 79.8]
  Week 18 | 77.7 [70.8 to 83.5] | 77.9 [71.1 to 83.7]
  Week 20 | 79.3 [72.7 to 85.0] | 76.2 [69.4 to 82.2]
  Week 24 | 79.9 [73.3 to 85.5] | 77.9 [71.1 to 83.7]
  Week 28 | 75.4 [68.4 to 81.5] | 77.9 [71.1 to 83.7]
  Week 32 | 77.1 [70.2 to 83.0] | 80.7 [74.1 to 86.1]
  Week 36 | 74.3 [67.2 to 80.5] | 80.7 [74.1 to 86.1]
  Week 40 | 74.9 [67.8 to 81.0] | 79.6 [72.9 to 85.2]
  Week 44 | 74.3 [67.2 to 80.5] | 80.7 [74.1 to 86.1]
  Week 48 | 76.0 [69.0 to 82.0] | 79.0 [72.3 to 84.7]
  Week 52 | 77.7 [70.8 to 83.5] | 79.0 [72.3 to 84.7]
  Week 56 | 77.7 [70.8 to 83.5] | 80.7 [74.1 to 86.1]
  Week 60 | 76.0 [69.0 to 82.0] | 79.0 [72.3 to 84.7]
  Week 64 | 78.2 [71.4 to 84.0] | 79.0 [72.3 to 84.7]
  Week 68 | 77.7 [70.8 to 83.5] | 76.8 [70.0 to 82.7]
  Week 72 | 79.9 [73.3 to 85.5] | 77.3 [70.6 to 83.2]
  Week 76 | 74.3 [67.2 to 80.5] | 77.3 [70.6 to 83.2]
  Week 80 | 74.3 [67.2 to 80.5] | 75.7 [68.8 to 81.7]
  Week 84 | 78.2 [71.4 to 84.0] | 73.5 [66.4 to 79.8]
  Week 88 | 77.7 [70.8 to 83.5] | 75.7 [68.8 to 81.7]
  Week 92 | 79.3 [72.7 to 85.0] | 74.0 [67.0 to 80.3]
  Week 96 | 78.8 [72.0 to 84.5] | 73.5 [66.4 to 79.8]
  Week 100 | 77.1 [70.2 to 83.0] | 73.5 [66.4 to 79.8]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 5 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 0.4, 95% CI 2-sided [-7.6 to 8.9]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 5 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 5.4, 95% CI 2-sided [-3.9 to 14.5]

14. Secondary Outcome: Percentage of Participants Who Gained >= 10 Letters in BCVA From Baseline or Reached BCVA >= 84 Letters at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 22.9 [17.0 to 29.8] | 23.8 [17.8 to 30.6]
  Week 6 | 34.6 [27.7 to 42.1] | 31.5 [24.8 to 38.8]
  Week 8 | 39.7 [32.4 to 47.2] | 36.5 [29.5 to 43.9]
  Week 12 | 43.0 [35.7 to 50.6] | 45.9 [39.4 to 53.4]
  Week 16 | 44.1 [36.7 to 51.7] | 49.7 [42.2 to 57.2]
  Week 18 | 47.5 [40.0 to 55.1] | 53.0 [45.5 to 60.5]
  Week 20 | 53.1 [45.5 to 60.6] | 56.9 [49.4 to 64.2]
  Week 24 | 56.4 [48.8 to 63.8] | 53.6 [46.0 to 61.0]
  Week 28 | 55.3 [47.7 to 62.7] | 55.2 [47.7 to 62.6]
  Week 32 | 58.7 [51.1 to 66.0] | 51.9 [44.4 to 59.4]
  Week 36 | 57.5 [49.9 to 64.9] | 55.2 [47.7 to 62.6]
  Week 40 | 58.1 [50.5 to 65.4] | 52.5 [44.9 to 59.9]
  Week 44 | 61.5 [53.9 to 68.6] | 56.9 [49.4 to 64.2]
  Week 48 | 60.9 [53.3 to 68.1] | 53.0 [45.5 to 60.5]
  Week 52 | 61.5 [53.9 to 68.6] | 58.6 [51.0 to 65.8]
  Week 56 | 62.0 [54.5 to 69.1] | 54.1 [46.6 to 61.6]
  Week 60 | 61.5 [53.9 to 68.6] | 54.7 [47.1 to 62.1]
  Week 64 | 63.7 [56.2 to 70.7] | 56.9 [49.4 to 64.2]
  Week 68 | 62.0 [54.5 to 69.1] | 57.5 [49.9 to 64.8]
  Week 72 | 63.7 [56.2 to 70.7] | 56.4 [48.8 to 63.7]
  Week 76 | 60.9 [53.3 to 68.1] | 56.9 [49.4 to 64.2]
  Week 80 | 57.5 [49.9 to 64.9] | 55.8 [48.2 to 63.2]
  Week 84 | 63.7 [56.2 to 70.7] | 58.6 [51.0 to 65.8]
  Week 88 | 61.5 [53.9 to 68.6] | 58.0 [50.5 to 65.3]
  Week 92 | 63.7 [56.2 to 70.7] | 58.6 [51.0 to 65.8]
  Week 96 | 62.6 [55.0 to 69.7] | 56.9 [49.4 to 64.2]
  Week 100 | 61.5 [53.9 to 68.6] | 54.1 [46.6 to 61.6]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 10 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 5.4, 95% CI 2-sided [-3.9 to 14.7]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 10 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 9.9, 95% CI 2-sided [-0.4 to 19.4]

15. Secondary Outcome: Percentage of Participants Who Gained >= 15 Letters in BCVA From Baseline or Reached BCVA >= 84 Letters at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 12.3 [7.9 to 18.0] | 9.4 [5.6 to 14.6]
  Week 6 | 13.4 [8.8 to 19.3] | 13.8 [9.1 to 19.7]
  Week 8 | 25.1 [19.0 to 32.2] | 16.0 [11.0 to 22.2]
  Week 12 | 25.1 [19.0 to 32.2] | 22.1 [16.3 to 28.9]
  Week 16 | 33.5 [26.7 to 40.9] | 25.4 [19.2 to 32.4]
  Week 18 | 31.8 [25.1 to 39.2] | 33.1 [26.3 to 40.5]
  Week 20 | 34.6 [27.7 to 42.1] | 32.6 [25.8 to 39.9]
  Week 24 | 41.9 [34.6 to 49.5] | 30.9 [24.3 to 38.2]
  Week 28 | 40.2 [33.0 to 47.8] | 37.0 [30.0 to 44.5]
  Week 32 | 44.1 [36.7 to 51.7] | 30.4 [23.8 to 37.6]
  Week 36 | 45.3 [37.8 to 52.8] | 32.6 [25.8 to 39.9]
  Week 40 | 44.7 [37.3 to 52.3] | 31.5 [24.8 to 38.8]
  Week 44 | 50.3 [42.7 to 57.8] | 35.4 [28.4 to 42.8]
  Week 48 | 41.9 [34.6 to 49.5] | 37.0 [30.0 to 44.5]
  Week 52 | 46.4 [38.9 to 54.0] | 37.6 [30.5 to 45.1]
  Week 56 | 46.4 [38.9 to 54.0] | 35.9 [28.9 to 43.4]
  Week 60 | 46.9 [39.4 to 54.5] | 38.7 [31.5 to 46.2]
  Week 64 | 50.3 [42.7 to 57.8] | 36.5 [29.5 to 43.9]
  Week 68 | 48.6 [41.1 to 56.2] | 35.9 [28.9 to 43.4]
  Week 72 | 48.0 [40.5 to 55.6] | 35.4 [28.4 to 42.8]
  Week 76 | 46.4 [38.9 to 54.0] | 40.9 [33.6 to 48.4]
  Week 80 | 43.6 [36.2 to 51.2] | 37.6 [30.5 to 45.1]
  Week 84 | 46.4 [38.9 to 54.0] | 37.0 [30.0 to 44.5]
  Week 88 | 47.5 [40.0 to 55.1] | 40.9 [33.6 to 48.4]
  Week 92 | 44.7 [37.3 to 52.3] | 40.3 [33.1 to 47.9]
  Week 96 | 46.9 [39.4 to 54.5] | 38.1 [31.0 to 45.6]
  Week 100 | 49.7 [42.2 to 57.3] | 37.6 [30.5 to 45.1]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 15 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 9.6, 95% CI 2-sided [-0.4 to 20.2]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Gain of >= 15 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 13.6, 95% CI 2-sided [3.3 to 23.5]

16. Secondary Outcome: Percentage of Participants Who Lost >= 5 ETDRS Letters in Best Corrected Visual Acuity (BCVA) From Baseline at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 3.4 [1.2 to 7.2] | 4.4 [1.9 to 8.5]
  Week 6 | 1.7 [0.3 to 4.8] | 3.3 [1.2 to 7.1]
  Week 8 | 1.1 [0.1 to 4.0] | 2.8 [0.9 to 6.3]
  Week 12 | 1.1 [0.1 to 4.0] | 2.2 [0.6 to 5.6]
  Week 16 | 0.6 [0.0 to 3.1] | 2.2 [0.6 to 5.6]
  Week 18 | 1.1 [0.1 to 4.0] | 1.1 [0.1 to 3.9]
  Week 20 | 2.2 [0.6 to 5.6] | 2.8 [0.9 to 6.3]
  Week 24 | 1.7 [0.3 to 4.8] | 3.3 [1.2 to 7.1]
  Week 28 | 1.7 [0.3 to 4.8] | 2.2 [0.6 to 5.6]
  Week 32 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 36 | 4.5 [1.9 to 8.6] | 1.1 [0.1 to 3.9]
  Week 40 | 3.9 [1.6 to 7.9] | 2.2 [0.6 to 5.6]
  Week 44 | 2.8 [0.9 to 6.4] | 2.2 [0.6 to 5.6]
  Week 48 | 2.8 [0.9 to 6.4] | 2.8 [0.9 to 6.3]
  Week 52 | 3.4 [1.2 to 7.2] | 3.3 [1.2 to 7.1]
  Week 56 | 5.0 [2.3 to 9.3] | 3.3 [1.2 to 7.1]
  Week 60 | 3.9 [1.6 to 7.9] | 4.4 [1.9 to 8.5]
  Week 64 | 2.8 [0.9 to 6.4] | 3.3 [1.2 to 7.1]
  Week 68 | 3.9 [1.6 to 7.9] | 2.8 [0.9 to 6.3]
  Week 72 | 4.5 [1.9 to 8.6] | 5.0 [2.3 to 9.2]
  Week 76 | 3.4 [1.2 to 7.2] | 4.4 [1.9 to 8.5]
  Week 80 | 2.8 [0.9 to 6.4] | 6.1 [3.1 to 10.6]
  Week 84 | 3.4 [1.2 to 7.2] | 7.7 [4.3 to 12.6]
  Week 88 | 3.9 [1.6 to 7.9] | 7.2 [3.9 to 12.0]
  Week 92 | 3.4 [1.2 to 7.2] | 6.6 [3.5 to 11.3]
  Week 96 | 3.9 [1.6 to 7.9] | 7.2 [3.9 to 12.0]
  Week 100 | 2.8 [0.9 to 6.4] | 8.3 [4.7 to 13.3]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 5 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.4, 95% CI 2-sided [-4.2 to 2.9]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 5 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -6.0, 95% CI 2-sided [-10.8 to -1.7]

17. Secondary Outcome: Percentage of Participants Who Lost >= 10 ETDRS Letters in Best Corrected Visual Acuity (BCVA) From Baseline at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | NA [NA to NA] — No participant satisfying the criteria of the response variable. | 1.1 [0.1 to 3.9]
  Week 6 | 1.1 [0.1 to 4.0] | 0.6 [0.0 to 3.0]
  Week 8 | 1.1 [0.1 to 4.0] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 12 | NA [NA to NA] — No participant satisfying the criteria of the response variable. | 0.6 [0.0 to 3.0]
  Week 16 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 18 | 1.1 [0.1 to 4.0] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 20 | 1.7 [0.3 to 4.8] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 24 | 1.7 [0.3 to 4.8] | 1.1 [0.1 to 3.9]
  Week 28 | 1.7 [0.3 to 4.8] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 32 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 36 | 3.4 [1.2 to 7.2] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 40 | 2.8 [0.9 to 6.4] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 44 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 48 | 2.2 [0.6 to 5.6] | 0.6 [0.0 to 3.0]
  Week 52 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 56 | 2.2 [0.6 to 5.6] | 1.1 [0.1 to 3.9]
  Week 60 | 1.7 [0.3 to 4.8] | 1.7 [0.3 to 4.8]
  Week 64 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 68 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 72 | 2.2 [0.6 to 5.6] | 1.7 [0.3 to 4.8]
  Week 76 | 2.2 [0.6 to 5.6] | 0.6 [0.0 to 3.0]
  Week 80 | 1.7 [0.3 to 4.8] | 1.7 [0.3 to 4.8]
  Week 84 | 2.2 [0.6 to 5.6] | 4.4 [1.9 to 8.5]
  Week 88 | 2.8 [0.9 to 6.4] | 3.9 [1.6 to 7.8]
  Week 92 | 2.8 [0.9 to 6.3] | 2.8 [0.9 to 6.3]
  Week 96 | 2.2 [0.6 to 5.6] | 3.9 [1.6 to 7.8]
  Week 100 | 2.2 [0.6 to 5.6] | 6.1 [3.1 to 10.6]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 10 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.2, 95% CI 2-sided [-3.2 to 2.4]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 10 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -4.1, 95% CI 2-sided [-8.4 to -0.1]

18. Secondary Outcome: Percentage of Participants Who Lost >= 15 ETDRS Letters in Best Corrected Visual Acuity (BCVA) From Baseline at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | NA [NA to NA] — No participant satisfying the criteria of the response variable. | 0.6 [0.0 to 3.0]
  Week 6 | 1.1 [0.1 to 4.0] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 8 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 12 | NA [NA to NA] — No participant satisfying the criteria of the response variable. | 0.6 [0.0 to 3.0]
  Week 16 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 18 | 1.1 [0.1 to 4.0] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 20 | 1.7 [0.3 to 4.8] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 24 | 1.1 [0.1 to 4.0] | 0.6 [0.0 to 3.0]
  Week 28 | 1.7 [0.3 to 4.8] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 32 | 1.7 [0.3 to 4.8] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 36 | 2.8 [0.9 to 6.4] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 40 | 2.2 [0.6 to 5.6] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 44 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 48 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 52 | 1.1 [0.1 to 4.0] | 1.7 [0.3 to 4.8]
  Week 56 | 1.7 [0.3 to 4.8] | 1.1 [0.1 to 3.9]
  Week 60 | 1.7 [0.3 to 4.8] | 1.7 [0.3 to 4.8]
  Week 64 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 68 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 72 | 2.2 [0.6 to 5.6] | 1.1 [0.1 to 3.9]
  Week 76 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 80 | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.0]
  Week 84 | 1.7 [0.3 to 4.8] | 2.2 [0.6 to 5.6]
  Week 88 | 1.7 [0.3 to 4.8] | 2.2 [0.6 to 5.6]
  Week 92 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 96 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 100 | 2.2 [0.6 to 5.6] | 3.3 [1.2 to 7.1]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 15 letters in BCVA at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.7, 95% CI 2-sided [-3.2 to 1.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Loss of >= 15 letters in BCVA at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -1.3, 95% CI 2-sided [-4.8 to 2.0]

19. Secondary Outcome: Percentage of Participants With an Absolute Best Corrected Visual Acuity (BCVA) >= 73 ETDRS Letters at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 55.3 [47.7 to 62.7] | 42.5 [35.2 to 50.1]
  Week 6 | 64.8 [57.3 to 71.8] | 49.7 [42.2 to 57.2]
  Week 8 | 66.5 [59.1 to 73.3] | 50.8 [43.3 to 58.3]
  Week 12 | 66.5 [59.1 to 73.3] | 59.7 [52.1 to 66.9]
  Week 16 | 69.8 [62.5 to 76.5] | 60.8 [53.3 to 67.9]
  Week 18 | 71.5 [64.3 to 78.0] | 64.6 [57.2 to 71.6]
  Week 20 | 71.5 [64.3 to 78.0] | 61.3 [53.8 to 68.5]
  Week 24 | 73.2 [66.1 to 79.5] | 60.2 [52.7 to 67.4]
  Week 28 | 72.6 [65.5 to 79.0] | 61.9 [54.4 to 69.0]
  Week 32 | 73.7 [66.7 to 80.0] | 59.1 [51.6 to 66.4]
  Week 36 | 70.4 [63.1 to 77.0] | 65.2 [57.8 to 72.1]
  Week 40 | 69.8 [62.5 to 76.5] | 60.2 [52.7 to 67.4]
  Week 44 | 73.7 [66.7 to 80.0] | 63.5 [56.1 to 70.5]
  Week 48 | 70.9 [63.7 to 77.5] | 61.3 [53.8 to 68.5]
  Week 52 | 73.7 [66.7 to 80.0] | 64.6 [57.2 to 71.6]
  Week 56 | 72.6 [65.5 to 79.0] | 66.9 [59.5 to 73.7]
  Week 60 | 70.9 [63.7 to 77.5] | 66.9 [59.5 to 73.7]
  Week 64 | 74.3 [67.2 to 80.5] | 68.5 [61.2 to 75.2]
  Week 68 | 71.5 [64.3 to 78.0] | 66.3 [58.9 to 73.1]
  Week 72 | 73.7 [66.7 to 80.0] | 65.2 [57.8 to 72.1]
  Week 76 | 72.6 [65.5 to 79.0] | 66.9 [59.5 to 73.7]
  Week 80 | 70.9 [63.7 to 77.5] | 64.1 [56.6 to 71.1]
  Week 84 | 70.9 [63.7 to 77.5] | 65.2 [57.8 to 72.1]
  Week 88 | 72.6 [65.5 to 79.0] | 63.5 [56.1 to 70.5]
  Week 92 | 71.5 [64.3 to 78.0] | 63.5 [56.1 to 70.5]
  Week 96 | 70.4 [63.1 to 77.0] | 62.4 [54.9 to 69.5]
  Week 100 | 70.9 [63.7 to 77.5] | 62.4 [54.9 to 69.5]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Absolute BCVA >= 73 letters at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 3.5, 95% CI 2-sided [-4.9 to 12.0]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Absolute BCVA >= 73 letters at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 3.6, 95% CI 2-sided [-5.4 to 12.6]

20. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CSFT) at Each Post-baseline Visit for the Study Eye
Description: The thickness of the retina was measured using Spectral Domain (SD) optical coherence tomography (OCT) equipment (SD-OCT) and reported as a difference, in micrometers. a negative change from baseline indicates a reduction in thickness, whereas a positive change from baseline indicates an increase. An increase in thickness may indicate a progression of the underlying disease. CSFT assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Micrometers
  Week 4: number analyzed (Participants) | 179 | 180
  Week 4 | -128.2 (131.47) | -113.9 (123.20)
  Week 6: number analyzed (Participants) | 179 | 180
  Week 6 | -136.9 (135.57) | -126.0 (124.82)
  Week 8: number analyzed (Participants) | 179 | 180
  Week 8 | -155.4 (139.09) | -130.8 (124.71)
  Week 12: number analyzed (Participants) | 179 | 180
  Week 12 | -160.8 (137.23) | -137.9 (132.30)
  Week 16: number analyzed (Participants) | 179 | 180
  Week 16 | -179.1 (137.26) | -145.3 (132.63)
  Week 18: number analyzed (Participants) | 179 | 180
  Week 18 | -175.8 (139.10) | -149.0 (132.28)
  Week 20: number analyzed (Participants) | 179 | 180
  Week 20 | -183.7 (139.76) | -151.0 (130.98)
  Week 24: number analyzed (Participants) | 179 | 180
  Week 24 | -183.3 (143.14) | -134.0 (136.67)
  Week 28: number analyzed (Participants) | 179 | 180
  Week 28 | -192.0 (145.85) | -161.4 (131.27)
  Week 32: number analyzed (Participants) | 179 | 180
  Week 32 | -178.6 (138.5) | -144.9 (135.93)
  Week 36: number analyzed (Participants) | 179 | 180
  Week 36 | -163.5 (144.34) | -162.9 (135.19)
  Week 40: number analyzed (Participants) | 179 | 180
  Week 40 | -183.3 (139.84) | -149.9 (132.66)
  Week 44: number analyzed (Participants) | 179 | 180
  Week 44 | -193.3 (144.12) | -163.5 (133.01)
  Week 48: number analyzed (Participants) | 179 | 180
  Week 48 | -172.8 (141.83) | -154.6 (130.54)
  Week 52: number analyzed (Participants) | 179 | 180
  Week 52 | -196.5 (144.44) | -165.0 (134.77)
  Week 56: number analyzed (Participants) | 179 | 180
  Week 56 | -191.08 (148.02) | -162.4 (132.53)
  Week 60: number analyzed (Participants) | 179 | 180
  Week 60 | -189.8 (147.93) | -166.2 (132.61)
  Week 64: number analyzed (Participants) | 179 | 180
  Week 64 | -193.2 (143.36) | -160.2 (137.83)
  Week 68: number analyzed (Participants) | 179 | 180
  Week 68 | -194.5 (141.47) | -169.8 (143.97)
  Week 72: number analyzed (Participants) | 179 | 180
  Week 72 | -190.4 (142.25) | -165.1 (141.38)
  Week 76: number analyzed (Participants) | 179 | 180
  Week 76 | -185.6 (143.68) | -174.7 (138.70)
  Week 80: number analyzed (Participants) | 179 | 180
  Week 80 | -185.7 (145.52) | -171.1 (138.53)
  Week 84: number analyzed (Participants) | 179 | 180
  Week 84 | -193.5 (142.53) | -175.1 (139.76)
  Week 88: number analyzed (Participants) | 179 | 180
  Week 88 | -191.0 (141.29) | -172.2 (138.08)
  Week 92: number analyzed (Participants) | 179 | 180
  Week 92 | -193.8 (142.07) | -180.1 (138.88)
  Week 96: number analyzed (Participants) | 179 | 180
  Week 96 | -197.2 (144.29) | -170.2 (154.37)
  Week 100: number analyzed (Participants) | 179 | 180
  Week 100 | -201.4 (142.90) | -173.9 (152.03)

21. Secondary Outcome: Average Mean Change From Baseline in Central Subfield Thickness (CSFT) Over the Period Week 40 Through Week 52 / Week 88 Through Week 100 for the Study Eye
Description: The thickness of the retina was measured using Spectral Domain (SD) optical coherence tomography (OCT) equipment (SD-OCT) and reported as a difference, in micrometers. a negative change from baseline indicates a reduction in thickness, whereas a positive change from baseline indicates an increase. An increase in thickness may indicate a progression of the underlying disease. CSFT assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment. For each participants, this endpoint was derived as the average of the changes from Baseline to Weeks 40, 44, 48, 52. Then the same was derived over the period Week 88 through Week 100, considering the average of the changes from Baseline to Weeks 88, 92, 96, 100. This endpoint was only assessed in the year-2 analysis (Week 100).
Time Frame: Baseline, period Week 40 through Week 52, period Week 88 through Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Micrometers
  period Week 40 through Week 52: number analyzed (Participants) | 179 | 180
  period Week 40 through Week 52 | -187.1 [-200.7 to -173.5] | -157.7 [-171.2 to -144.1]
  period Week 88 through Week 100: number analyzed (Participants) | 179 | 180
  period Week 88 through Week 100 | -196.6 [-210.9 to -182.3] | -173.4 [-187.6 to -159.1]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT over period Week 40 through Week 52; Test type: Other — Treatment difference; p < 0.003, ANOVA; LS mean difference = -29.4, 95% CI 2-sided [-48.6 to -10.2], Standard Error of Mean 9.76
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT over period Week 40 through Week 52; Test type: Superiority; p = 0.001, ANOVA
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT over period Week 88 through Week 100; Test type: Other — Treatment difference; LS mean difference = -23.2, 95% CI 2-sided [-43.5 to -3.0], Standard Error of Mean 10.28

22. Secondary Outcome: Average Mean Change From Baseline in CSFT Over the Period Week 4 to Week 52 / 100 for the Study Eye
Description: as for outcome 20
Time Frame: Baseline, period Week 4 through Week 52, period Week 4 through Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: Micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Micrometers
  period Week 4 through Week 52 | -172.8 [-185.8 to -159.8] | -145.4 [-158.4 to -132.4]
  period Week 4 through Week 100: number analyzed (Participants) | 179 | 180
  period Week 4 through Week 100 | -181.8 [-194.7 to -168.9] | -156.1 [-169.0 to -143.2]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT over period Week 4 through Week 52; Test type: Other — Treatment difference; LS mean difference = -27.4, 95% CI 2-sided [-45.8 to -9.0], Standard Error of Mean 9.35
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT over period Week 4 through Week 100; Test type: Other — Treatment difference; LS mean difference = -25.8, 95% CI 2-sided [-44.0 to -7.5], Standard Error of Mean 9.29

23. Secondary Outcome: Percentage of Participants With Normal CSFT Thickness (<280 Micrometers) at Each Post-baseline Visit for the Study Eye
Description: The thickness of the retina was measured using Spectral Domain (SD) optical coherence tomography (OCT) equipment (SD-OCT) and reported as a difference, in micrometers. CSFT assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: as for outcome 9
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 12.8 [8.3 to 18.7] | 13.3 [8.7 to 19.2]
  Week 6 | 16.8 [11.6 to 23.1] | 14.4 [9.7 to 20.4]
  Week 8 | 22.9 [17.0 to 29.8] | 16.7 [11.5 to 22.9]
  Week 12 | 30.2 [23.5 to 37.5] | 24.4 [18.4 to 31.4]
  Week 16 | 36.9 [29.8 to 44.4] | 29.4 [22.9 to 36.7]
  Week 18 | 39.1 [31.9 to 46.7] | 30.0 [23.4 to 37.3]
  Week 20 | 42.5 [35.1 to 50.1] | 31.1 [24.4 to 38.4]
  Week 24 | 48.6 [41.1 to 56.2] | 29.4 [22.9 to 36.7]
  Week 28 | 50.3 [42.7 to 57.8] | 33.9 [27.0 to 41.3]
  Week 32 | 48.0 [40.5 to 55.6] | 30.6 [23.9 to 37.8]
  Week 36 | 38.5 [31.4 to 46.1] | 38.9 [31.7 to 46.4]
  Week 40 | 51.4 [43.8 to 58.9] | 37.2 [30.1 to 44.7]
  Week 44 | 51.4 [43.8 to 58.9] | 38.9 [31.7 to 46.4]
  Week 48 | 49.7 [42.2 to 57.3] | 37.2 [30.1 to 44.7]
  Week 52 | 57.5 [49.9 to 64.9] | 41.4 [34.2 to 49.0]
  Week 56 | 57.5 [49.9 to 64.9] | 40.3 [33.1 to 47.9]
  Week 60 | 53.1 [45.5 to 60.6] | 40.3 [33.1 to 47.9]
  Week 64 | 54.2 [46.6 to 61.6] | 38.1 [31.0 to 45.6]
  Week 68 | 53.6 [46.0 to 61.1] | 41.4 [34.2 to 49.0]
  Week 72 | 56.4 [48.8 to 63.8] | 38.7 [31.5 to 46.2]
  Week 76 | 55.3 [47.7 to 62.7] | 42.5 [35.2 to 50.1]
  Week 80 | 57.0 [49.4 to 64.3] | 39.8 [32.6 to 47.3]
  Week 84 | 57.0 [49.4 to 64.3] | 43.1 [35.8 to 50.6]
  Week 88 | 56.4 [48.8 to 63.8] | 41.4 [34.2 to 49.0]
  Week 92 | 57.0 [49.4 to 64.3] | 45.9 [38.4 to 53.4]
  Week 96 | 59.8 [52.2 to 67.0] | 43.6 [36.3 to 51.2]
  Week 100 | 62.0 [54.5 to 69.1] | 47.0 [39.5 to 54.5]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT thickness (<280 micrometers) at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 16.3, 95% CI 2-sided [5.7 to 25.9]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; CSFT thickness (<280 micrometers) at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 14.7, 95% CI 2-sided [4.2 to 24.9]

24. Secondary Outcome: Percentage of Patients With Presence of Subretinal Fluid (SRF) in the Study Eye at Each Post-baseline Visit
Description: Presence of Subretinal Fluid (SRF) in the study eye was assessed by spectral domain optical coherence tomography (SD-OCT), angiography, and/or color fundus photography. Subretinal fluid status assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Week 4, Week 6, Week 8, Week 12, Week 16, Week 18, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56, Week 60, Week 64, Week 68, Week 72, Week 76, Week 80, Week 84, Week 88, Week 92, Week 96, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 12.3 [7.9 to 18.0] | 19.3 [13.9 to 25.9]
  Week 6 | 10.1 [6.1 to 15.4] | 13.8 [9.1 to 19.7]
  Week 8 | 5.6 [2.7 to 10.0] | 12.2 [7.8 to 17.8]
  Week 12 | 3.9 [1.6 to 7.9] | 7.7 [4.3 to 12.6]
  Week 16 | 1.7 [0.3 to 4.8] | 3.9 [1.6 to 7.8]
  Week 18 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 20 | 1.7 [0.3 to 4.8] | 3.3 [1.2 to 7.1]
  Week 24 | 2.2 [0.6 to 5.6] | 6.6 [3.5 to 11.3]
  Week 28 | 2.2 [0.6 to 5.6] | 2.8 [0.9 to 6.3]
  Week 32 | 5.0 [2.3 to 9.3] | 3.9 [1.6 to 7.8]
  Week 36 | 6.7 [3.5 to 11.4] | 1.7 [0.3 to 4.8]
  Week 40 | 4.5 [1.9 to 8.6] | 2.8 [0.9 to 6.3]
  Week 44 | 2.2 [0.6 to 5.6] | 2.8 [0.9 to 6.3]
  Week 48 | 6.1 [3.1 to 10.7] | 5.0 [2.3 to 9.2]
  Week 52 | 1.7 [0.3 to 4.8] | 3.3 [1.2 to 7.1]
  Week 56 | 2.8 [0.9 to 6.4] | 2.2 [0.6 to 5.6]
  Week 60 | 2.8 [0.9 to 6.4] | 2.2 [0.6 to 5.6]
  Week 64 | 2.2 [0.6 to 5.6] | 3.9 [1.6 to 7.8]
  Week 68 | 3.4 [1.2 to 7.2] | 4.4 [1.9 to 8.5]
  Week 72 | 3.4 [1.2 to 7.2] | 2.8 [0.9 to 6.3]
  Week 76 | 3.9 [1.6 to 7.9] | 2.2 [0.6 to 5.6]
  Week 80 | 4.5 [1.9 to 8.6] | 2.2 [0.6 to 5.6]
  Week 84 | 2.2 [0.6 to 5.6] | 2.2 [0.6 to 5.6]
  Week 88 | 3.4 [1.2 to 7.2] | 2.2 [0.6 to 5.6]
  Week 92 | 1.7 [0.3 to 4.8] | 1.1 [0.1 to 3.9]
  Week 96 | 2.2 [0.6 to 5.6] | 2.8 [0.9 to 6.3]
  Week 100 | 2.2 [0.6 to 5.6] | 2.8 [0.9 to 6.3]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Subretinal Fluid (SRF) at Week 52; Test type: Other; Clopper-Pearson exact method = -1.2, 95% CI 2-sided [-4.5 to 2.1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Subretinal Fluid (SRF) at Week 100; Test type: Other — Treatment Difference; Clopper-Pearson exact method = -0.2, 95% CI 2-sided [-3.4 to 3.4]

25. Secondary Outcome: Percentage of Patients With Presence of Intraretinal Fluid (IRF) in the Study Eye at Each Post-baseline Visit
Description: Presence of Intraretinal Fluid (IRF) in the study eye was assessed by spectral domain optical coherence tomography (SD-OCT), angiography, and/or color fundus photography. Intraretinal fluid status assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: as for outcome 24
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 88.3 [82.6 to 92.6] | 89.0 [83.5 to 93.1]
  Week 6 | 85.5 [79.4 to 90.3] | 86.2 [80.3 to 90.9]
  Week 8 | 87.2 [81.3 to 91.7] | 84.5 [78.4 to 89.5]
  Week 12 | 83.8 [77.6 to 88.9] | 85.6 [79.7 to 90.4]
  Week 16 | 76.0 [69.0 to 82.0] | 84.0 [77.8 to 89.0]
  Week 18 | 77.7 [70.8 to 83.5] | 81.2 [74.8 to 86.6]
  Week 20 | 72.6 [65.5 to 79.0] | 79.6 [72.9 to 85.2]
  Week 24 | 69.8 [62.5 to 76.5] | 82.3 [76.0 to 87.6]
  Week 28 | 67.6 [60.2 to 74.4] | 75.1 [68.2 to 81.3]
  Week 32 | 67.6 [60.2 to 74.4] | 76.8 [70.0 to 82.7]
  Week 36 | 73.2 [66.1 to 79.5] | 72.4 [65.3 to 78.7]
  Week 40 | 57.5 [49.9 to 64.9] | 74.0 [67.0 to 80.3]
  Week 44 | 56.4 [48.8 to 63.8] | 71.3 [64.1 to 77.7]
  Week 48 | 60.9 [53.3 to 68.1] | 75.7 [68.8 to 81.7]
  Week 52 | 53.6 [46.0 to 61.1] | 72.9 [65.8 to 79.3]
  Week 56 | 51.4 [43.8 to 58.9] | 70.2 [62.9 to 76.7]
  Week 60 | 55.3 [47.7 to 62.7] | 69.1 [61.8 to 75.7]
  Week 64 | 48.6 [41.1 to 56.2] | 69.6 [62.4 to 76.2]
  Week 68 | 47.5 [40.0 to 55.1] | 66.9 [59.5 to 73.7]
  Week 72 | 45.8 [38.4 to 53.4] | 66.9 [59.5 to 73.7]
  Week 76 | 50.3 [42.7 to 57.8] | 63.0 [55.5 to 70.0]
  Week 80 | 45.8 [38.4 to 53.4] | 65.7 [58.3 to 72.6]
  Week 84 | 40.2 [33.0 to 47.8] | 63.0 [55.5 to 70.0]
  Week 88 | 48.0 [40.5 to 55.6] | 64.1 [56.6 to 71.1]
  Week 92 | 44.7 [37.3 to 52.3] | 59.1 [51.6 to 66.4]
  Week 96 | 41.3 [34.0 to 48.9] | 61.9 [54.4 to 69.0]
  Week 100 | 40.8 [33.5 to 48.4] | 56.9 [49.4 to 64.2]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Intraretinal Fluid (IRF) at Week 52; Test type: Other — Treatment Difference; Clopper-Pearson exact method = -19.1, 95% CI 2-sided [-28.9 to -9.2]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Intraretinal Fluid (IRF) at Week 100; Test type: Other — Treatment Difference; Clopper-Pearson exact method = -16.1, 95% CI 2-sided [-26.3 to -5.7]

26. Secondary Outcome: Percentage of Patients With Presence of Subretinal Fluid (SRF) and/or Intraretinal Fluid (IRF) in the Study Eye at Each Post-baseline Visit
Description: Presence of Subretinal Fluid (SRF) and/or Intraretinal Fluid (IRF) in the study eye was assessed by spectral domain optical coherence tomography (SD-OCT), angiography, and/or color fundus photography. Fluid status (SRF and/or IRF) assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: as for outcome 24
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 4 | 90.5 [85.2 to 94.4] | 90.6 [85.4 to 94.4]
  Week 6 | 86.6 [80.7 to 91.2] | 88.4 [82.8 to 92.7]
  Week 8 | 87.2 [81.3 to 91.7] | 85.6 [79.7 to 90.4]
  Week 12 | 83.8 [77.6 to 88.9] | 86.2 [80.3 to 90.9]
  Week 16 | 76.0 [69.0 to 82.0] | 84.0 [77.8 to 89.0]
  Week 18 | 78.2 [71.4 to 84.0] | 81.2 [74.8 to 86.6]
  Week 20 | 73.2 [66.1 to 79.5] | 79.6 [72.9 to 85.2]
  Week 24 | 70.4 [63.1 to 77.0] | 82.3 [76.0 to 87.6]
  Week 28 | 68.7 [61.4 to 75.4] | 75.1 [68.2 to 81.3]
  Week 32 | 68.7 [61.4 to 75.4] | 76.8 [70.0 to 82.7]
  Week 36 | 73.7 [66.7 to 80.0] | 72.4 [65.3 to 78.7]
  Week 40 | 58.1 [50.5 to 65.4] | 74.0 [67.0 to 80.3]
  Week 44 | 57.0 [49.4 to 64.3] | 71.3 [64.1 to 77.7]
  Week 48 | 61.5 [53.9 to 68.6] | 75.7 [68.8 to 81.7]
  Week 52 | 54.2 [46.6 to 61.6] | 72.9 [65.8 to 79.3]
  Week 56 | 52.0 [44.4 to 59.5] | 70.2 [62.9 to 76.7]
  Week 60 | 55.3 [47.7 to 62.7] | 69.1 [61.8 to 75.7]
  Week 64 | 49.2 [41.6 to 56.7] | 69.6 [62.4 to 76.2]
  Week 68 | 48.0 [40.5 to 55.6] | 68.0 [60.6 to 74.7]
  Week 72 | 46.9 [39.4 to 54.5] | 66.9 [59.5 to 73.7]
  Week 76 | 50.8 [43.3 to 58.4] | 63.0 [55.5 to 70.0]
  Week 80 | 46.4 [38.9 to 54.0] | 65.7 [58.3 to 72.6]
  Week 84 | 40.8 [33.5 to 48.4] | 63.0 [55.5 to 70.0]
  Week 88 | 48.6 [41.1 to 56.2] | 64.1 [56.6 to 71.1]
  Week 92 | 45.3 [37.8 to 52.8] | 59.1 [51.6 to 66.4]
  Week 96 | 41.3 [34.0 to 48.9] | 61.9 [54.4 to 69.0]
  Week 100 | 40.8 [33.5 to 48.4] | 56.9 [49.4 to 64.2]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Subretinal Fluid (SRF) and/or Intraretinal Fluid (IRF) at Week 52; Test type: Other — Treatment Difference; Clopper-Pearson exact method = -18.4, 95% CI 2-sided [-28.5 to -8.3]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Subretinal Fluid (SRF) and/or Intraretinal Fluid (IRF) at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -16.2, 95% CI 2-sided [-26.4 to -5.9]

27. Secondary Outcome: Percentage of Participants With Presence of Leakage on Fluorescein Angiography (FA) at Weeks 52 and 100
Description: Presence of leakage on Fluorescein Angiography as assessed by fluorescein angiography. Leakage on FA assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Week 52, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 52 | 54.7 [47.2 to 62.2] | 79.4 [72.8 to 85.1]
  Week 100 | 46.9 [39.4 to 54.5] | 65.6 [58.1 to 72.5]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Fluorescein Angiography (FA) at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = -25.4, 95% CI 2-sided [-34.4 to -16.3]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Fluorescein Angiography (FA) at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -19.1, 95% CI 2-sided [-29.1 to -8.2]

28. Secondary Outcome: Percentage of Participants With With >=2-step Improvement From Baseline in ETDRS Diabetic Retinopathy Severity Scale (ETDRS-DRSS) Score
Description: The Diabetic Retinopathy Disease Severity Scale measures the 5 levels of diabetic retinopathy - none, mild, moderate, severe, and proliferative. DRSS assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 28 | 25.0 [18.8 to 32.1] | 20.9 [15.2 to 27.6]
  Week 52 | 29.0 [22.4 to 36.3] | 27.7 [21.2 to 34.9]
  Week 76 | 30.1 [23.4 to 37.5] | 30.5 [23.8 to 37.9]
  Week 100 | 35.8 [28.7 to 43.4] | 31.1 [24.3 to 38.5]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=2-step improvement in ETDRS-DRSS at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 1.1, 95% CI 2-sided [-5.6 to 7.8]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=2-step improvement in ETDRS-DRSS at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 4.5, 95% CI 2-sided [-1.7 to 10.8]

29. Secondary Outcome: Percentage of Participants With With >=3-step Improvement From Baseline in ETDRS Diabetic Retinopathy Severity Scale (ETDRS-DRSS) Score
Description: as for outcome 28
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 28 | 13.1 [8.5 to 19.0] | 11.3 [7.0 to 16.9]
  Week 52 | 14.8 [9.9 to 20.9] | 15.3 [10.3 to 21.4]
  Week 76 | 18.8 [13.3 to 25.3] | 15.3 [10.3 to 21.4]
  Week 100 | 21.0 [15.3 to 27.8] | 16.9 [11.7 to 23.3]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=3-step improvement in ETDRS-DRSS at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.6, 95% CI 2-sided [-7.1 to 5.7]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=3-step improvement in ETDRS-DRSS at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 3.9, 95% CI 2-sided [-2.3 to 10.0]

30. Secondary Outcome: Percentage of Participants With With >=2-step Worsening From Baseline in ETDRS Diabetic Retinopathy Severity Scale (ETDRS-DRSS) Score
Description: The Diabetic Retinopathy Disease Severity Scale was based on 7-field stereo color fundus photography and measured 5 levels of diabetic retinopathy - none, mild, moderate, severe, and proliferative. DRSS assessments after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and replaced by the last value prior to start of this alternative treatment.
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 28 | 2.3 [0.6 to 5.7] | 0.6 [0.0 to 3.1]
  Week 52 | 1.7 [0.4 to 4.9] | 0.6 [0.0 to 3.1]
  Week 76 | 3.4 [1.3 to 7.3] | 0.6 [0.0 to 3.1]
  Week 100 | 4.5 [2.0 to 8.8] | 1.7 [0.4 to 4.9]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=2-step worsening in ETDRS-DRSS at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 1.1, 95% CI 2-sided [-1.0 to 3.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=2-step worsening in ETDRS-DRSS at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = 2.9, 95% CI 2-sided [-0.5 to 6.9]

31. Secondary Outcome: Percentage of Participants With With >=3-step Worsening From Baseline in ETDRS Diabetic Retinopathy Severity Scale (ETDRS-DRSS) Score
Description: as for outcome 30
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants
  Week 28 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 52 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 76 | 0.6 [0.0 to 3.1] | NA [NA to NA] — No participant satisfying the criteria of the response variable.
  Week 100 | 0.6 [0.0 to 3.1] | 1.1 [0.1 to 4.0]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=3-step worsening in ETDRS-DRSS at Week 52; Test type: Other — Treatment difference; Clopper-Pearson exact method = 0.6, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; >=3-step worsening in ETDRS-DRSS at Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.6, 95% CI 2-sided [-2.6 to 1.3]

32. Secondary Outcome: Percentage of Participants With Progression to Proliferative Diabetic Retinopathy (PDR) as Assessed by ETDRS-DRSS Score of at Least 61 by Week 100
Description: as for outcome 30
Time Frame: Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Percentage of Participants | 0.6 [0.0 to 3.4] | 0.6 [0.0 to 3.4]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proliferative diabetic retinopathy (PDR) of at least 61 by Week 100; Test type: Other — Treatment difference; Clopper-Pearson exact method = -0.0, 95% CI 2-sided [-2.1 to 1.9]

33. Secondary Outcome: Number of Participants With Ocular and Non-ocular Adverse Events (AEs)
Description: The number of participants with ocular and non-ocular adverse events was was assessed by CTCAE and reported categorically: Mild, Moderate, Severe.
Time Frame: From randomization till 30 days safety follow-up, assessed up to 35 months.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Participants
  Ocular adverse events: number analyzed (Participants) | 73 | 74
  Ocular adverse events: Mild | 52 | 47
  Ocular adverse events: Moderate | 15 | 23
  Ocular adverse events: Severe | 6 | 4
  Non-ocular adverse events: number analyzed (Participants) | 136 | 141
  Non-ocular adverse events: Mild | 52 | 51
  Non-ocular adverse events: Moderate | 51 | 50
  Non-ocular adverse events: Severe | 33 | 40

34. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Composite Score
Description: The survey consisted of 25 items representing 11 vision related constructs (general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, peripheral vision) plus a single-item general health rating question. The score of each individual question ranged from 0 (worst) to 100 which indicated the best possible response. The composite score and score of each construct also ranged from 0 to 100 as they were calculated as total scores divided by the number of questions. The higher the values of total scores represented better outcome.
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: Full Analysis Set - Observed. Data after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 5.7 (11.91) | 6.3 (10.19)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 8.9 (11.67) | 6.7 (12.12)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 9.8 (12.22) | 7.6 (11.81)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 9.0 (12.94) | 6.2 (14.13)

35. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - General Vision
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 9.0 (16.11) | 10.2 (15.63)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 11.2 (17.05) | 10.5 (17.14)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 12.4 (16.49) | 12.0 (16.40)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 12.0 (16.25) | 10.1 (18.73)

36. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Ocular Pain
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 4.1 (19.52) | 4.6 (18.48)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 4.6 (18.75) | 4.4 (17.92)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 6.2 (16.95) | 4.6 (18.68)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 4.3 (16.60) | 5.4 (20.77)

37. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Near Activities
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 165 | 168
  Week 28 | 6.4 (20.83) | 6.3 (18.42)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 10.5 (20.30) | 9.3 (19.57)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 11.0 (21.91) | 9.2 (18.76)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 13.0 (20.21) | 7.3 (21.71)

38. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Distance Activities
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 6.2 (18.87) | 5.6 (15.78)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 11.7 (17.62) | 8.2 (17.12)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 12.1 (18.32) | 8.1 (16.71)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 11.4 (18.94) | 6.6 (19.07)

39. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Social Functioning
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 3.3 (15.82) | 4.4 (16.48)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 7.1 (16.22) | 4.9 (15.59)
  Week 76: number analyzed (Participants) | 131 | 145
  Week 76 | 6.3 (16.65) | 5.0 (15.34)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 6.1 (16.78) | 4.1 (17.55)

40. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Mental Health
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 7.9 (19.53) | 10.1 (19.90)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 12.6 (22.42) | 10.1 (22.78)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 13.5 (21.02) | 13.1 (23.10)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 13.3 (20.91) | 11.6 (26.31)

41. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Role Difficulties
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 6.9 (25.13) | 9.4 (23.41)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 12.2 (24.76) | 8.7 (27.21)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 14.0 (28.44) | 11.4 (27.83)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 12.3 (28.14) | 10.2 (27.12)

42. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Dependency
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 5.5 (19.39) | 3.6 (20.34)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 7.6 (19.53) | 3.9 (22.49)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 7.3 (20.19) | 5.6 (23.24)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 6.8 (19.85) | 2.9 (24.79)

43. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Driving
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 94 | 87
  Week 28 | 1.4 (18.75) | 4.8 (12.24)
  Week 52: number analyzed (Participants) | 84 | 76
  Week 52 | 6.4 (14.63) | 4.2 (12.81)
  Week 76: number analyzed (Participants) | 72 | 74
  Week 76 | 8.9 (15.95) | 2.8 (15.88)
  Week 100: number analyzed (Participants) | 78 | 74
  Week 100 | 5.4 (15.81) | 1.2 (16.75)

44. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Color Vision
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 165 | 166
  Week 28 | 3.5 (15.10) | 4.2 (12.50)
  Week 52: number analyzed (Participants) | 142 | 147
  Week 52 | 5.8 (15.08) | 3.6 (13.09)
  Week 76: number analyzed (Participants) | 131 | 141
  Week 76 | 5.2 (15.73) | 3.9 (13.79)
  Week 100: number analyzed (Participants) | 129 | 141
  Week 100 | 4.3 (14.70) | 3.2 (15.48)

45. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): Subscale Score - Peripheral Vision
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 167
  Week 28 | 5.3 (18.83) | 4.0 (16.99)
  Week 52: number analyzed (Participants) | 143 | 149
  Week 52 | 7.2 (18.68) | 3.2 (19.77)
  Week 76: number analyzed (Participants) | 132 | 144
  Week 76 | 9.3 (19.64) | 4.3 (17.82)
  Week 100: number analyzed (Participants) | 130 | 144
  Week 100 | 8.5 (19.33) | 2.3 (19.37)

46. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25): General Health Rating
Description: as for outcome 34
Time Frame: Baseline, Week 28, Week 52, Week 76, Week 100
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 181
Score on a scale
  Week 28: number analyzed (Participants) | 166 | 168
  Week 28 | 3.9 (18.66) | 4.3 (19.92)
  Week 52: number analyzed (Participants) | 143 | 150
  Week 52 | 5.8 (22.34) | 4.8 (23.12)
  Week 76: number analyzed (Participants) | 132 | 145
  Week 76 | 8.9 (21.21) | 7.1 (22.57)
  Week 100: number analyzed (Participants) | 130 | 145
  Week 100 | 6.7 (19.14) | 5.7 (21.80)

47. Secondary Outcome: Systemic Brolucizumab Concentration
Description: Serum samples were taken approximately 24 hours after the first dose and 24 hours after the treatment at Week 24 to confirm the systemic brolucizumab exposure in patients with visual impairment due to diabetic macular edema.
Time Frame: Up to Week 24
Population: Safety Set. Data after start of alternative diabetic macular edema (DME) treatment in the study eye were censored and not included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
ng/mL
  Day 2: number analyzed (Participants) | 28 | 0
  Day 2 | 56.2 (10.4) |
  Week 4: number analyzed (Participants) | 162 | 0
  Week 4 | 0.760 (1.98) |
  Week 12: number analyzed (Participants) | 168 | 0
  Week 12 | NA (NA) — NA = not estimable: Below the limit of quantitation (<0.5 ng/mL) |
  Week 24: number analyzed (Participants) | 165 | 0
  Week 24 | NA (NA) — NA = not estimable: Below the limit of quantitation (<0.5 ng/mL) |
  Week 24 + 1 Day: number analyzed (Participants) | 21 | 0
  Week 24 + 1 Day | 41.5 (80.5) |

48. Secondary Outcome: Distribution of Integrated Anti-Drug Antibody (ADA) Status in the Brolucizumab Arm
Description: Integrated ADA Status was categorized: ADA negative or ADA positive with no boost, Induced or Boosted, Missing ADA at pre-dose or no post-dose ADA data.
  * ADA negative: (a) ADA negative at all time points (pre-dose and post-dose), (b) ADA negative at pre-dose and no titer values above 40 at all other time points, (c) ADA titer of 40 at pre-dose but negative at all other time points.
  * ADA positive with no boost: ADA positive at pre-dose, post-dose titer values do not increase from pre-dose by more than 3-fold (1 dilution) at any time point.
  * Induced: ADA negative at pre-dose, post-dose titer value of 120 or more at any time point.
  * Boosted: ADA positive at pre-dose, post-dose titer values increase from pre-dose by more than 3-fold (1 dilution) at any time point.
Time Frame: Up to Week 100
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
Participants
  ADA negative or ADA positive with no boost | 146 |
  Induced or Boosted | 27 |
  Missing ADA at pre-dose or no post-dose ADA data | 6 |

49. Secondary Outcome: Distribution of Integrated Anti-Drug Antibody (ADA) Status in the Brolucizumab Arm - Adjusted for Pre-existing ADA Status
Description: Integrated ADA Status - adjusted for pre-existing ADA status was categorized: ADA negative, ADA positive with no boost, Induced, Boosted.
  * ADA negative: (a) ADA negative at all time points (pre-dose and post-dose), (b) ADA negative at pre-dose and no titer values above 40 at all other time points, (c) ADA titer of 40 at pre-dose but negative at all other time points.
  * ADA positive with no boost: ADA positive at pre-dose, post-dose titer values do not increase from pre-dose by more than 3-fold (1 dilution) at any time point.
  * Induced: ADA negative at pre-dose, post-dose titer value of 120 or more at any time point.
  * Boosted: ADA positive at pre-dose, post-dose titer values increase from pre-dose by more than 3-fold (1 dilution) at any time point.
Time Frame: Up to Week 100
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
Participants
  ADA negative/ADA Negative or titer value of 40 at pre-dose: number analyzed (Participants) | 84 | 0
  ADA negative/ADA Negative or titer value of 40 at pre-dose | 53 |
  ADA positive with no boost/ADA Positive at pre-dose: number analyzed (Participants) | 110 | 0
  ADA positive with no boost/ADA Positive at pre-dose | 93 |
  Induced/ADA Negative at pre-dose: number analyzed (Participants) | 64 | 0
  Induced/ADA Negative at pre-dose | 14 |
  Boosted/ADA Positive at pre-dose: number analyzed (Participants) | 110 | 0
  Boosted/ADA Positive at pre-dose | 13 |

50. Secondary Outcome: Pre-existing ADA Status and Incidence of Adverse Event of Special Interest (AESI) in the Study Eye
Description: Pre-existing ADA status and incidence of Adverse Event of Special Interest (AESI) in the study eye was categorized: Negative, Positive.
Time Frame: Up to Week 100
Population: Safety Set. AEs started after the subject discontinued study treatment and started alternative diabetic macular edema (DME) treatment in the study eye were censored and not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
Participants
  Negative: number analyzed (Participants) | 64 | 0
  Negative: At least 1 AESI | 1 |
  Negative: No AESI | 63 |
  Postive: number analyzed (Participants) | 110 | 0
  Postive: At least 1 AESI | 5 |
  Postive: No AESI | 105 |

51. Secondary Outcome: Integrated ADA Status up to Week 100 and Incidence of Adverse Event of Special Interest (AESI) in the Study Eye.
Description: Integrated ADA status up to Week 100 and incidence of Adverse Event of Special Interest (AESI) in the study eye was categorized: ADA-negative or no boost, Induced or boosted.
Time Frame: Up to Week 100
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 179 | 0
Participants
  ADA-negative or no boost: number analyzed (Participants) | 146 | 0
  ADA-negative or no boost: At least 1 AESI | 4 |
  ADA-negative or no boost: No AESI | 142 |
  Induced or boosted: number analyzed (Participants) | 27 | 0
  Induced or boosted: At least 1 AESI | 2 |
  Induced or boosted: No AESI | 25 |

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days after last dose (maximum 35 months)
Description: Adverse Events (AEs) and All-cause mortality were collected in the Safety Set
Groups:
- Brolucizumab 6mg: Brolucizumab 6 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule
- Aflibercept 2mg: Aflibercept 2 mg/0.05 mL, as labeled, 5 loading doses, with subsequent doses every 8 weeks
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 13/179 | 9/181 | 22/360
Serious Adverse Events (participants affected / at risk) | 53/179 | 60/181 | 113/360
Other Adverse Events (participants affected / at risk) | 131/179 | 134/181 | 265/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=179) | Aflibercept 2mg (N=181) | Overall (N=360)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 2
Angina pectoris (Cardiac disorders) | 2 | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 2
Cardiac failure (Cardiac disorders) | 2 | 4 | 6
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1 | 2
Coronary artery disease (Cardiac disorders) | 1 | 2 | 3
Coronary artery stenosis (Cardiac disorders) | 2 | 1 | 3
Myocardial infarction (Cardiac disorders) | 0 | 3 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 1 | 1
Glaucoma - Study eye (Eye disorders) | 1 | 0 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 1 | 0 | 1
Retinal detachment - Study eye (Eye disorders) | 0 | 1 | 1
Retinal tear - Study eye (Eye disorders) | 0 | 1 | 1
Uveitis - Fellow eye (Eye disorders) | 0 | 1 | 1
Uveitis - Study eye (Eye disorders) | 1 | 1 | 2
Vitreous haemorrhage - Fellow eye (Eye disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2
Death (General disorders) | 1 | 2 | 3
Mass (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 4 | 3 | 7
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1
Endophthalmitis - Study eye (Infections and infestations) | 2 | 1 | 3
Erysipelas (Infections and infestations) | 1 | 1 | 2
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 3 | 2 | 5
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 1
Ophthalmic herpes zoster - Study eye (Infections and infestations) | 1 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 3 | 7
Pneumonia viral (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Streptococcal infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Arachnoiditis (Nervous system disorders) | 0 | 1 | 1
Bickerstaff's encephalitis (Nervous system disorders) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebellar stroke (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 4
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 3 | 3
Diabetic nephropathy (Renal and urinary disorders) | 1 | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Breast hypoplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=179) | Aflibercept 2mg (N=181) | Overall (N=360)
Anaemia (Blood and lymphatic system disorders) | 8 | 8 | 16
Blepharitis - Fellow eye (Eye disorders) | 2 | 5 | 7
Blepharitis - Study eye (Eye disorders) | 2 | 4 | 6
Cataract - Fellow eye (Eye disorders) | 11 | 16 | 27
Cataract - Study eye (Eye disorders) | 12 | 19 | 31
Conjunctival haemorrhage - Fellow eye (Eye disorders) | 1 | 9 | 10
Conjunctival haemorrhage - Study eye (Eye disorders) | 9 | 6 | 15
Diabetic retinal oedema - Fellow eye (Eye disorders) | 18 | 16 | 34
Diabetic retinopathy - Fellow eye (Eye disorders) | 5 | 1 | 6
Dry eye - Fellow eye (Eye disorders) | 9 | 7 | 16
Dry eye - Study eye (Eye disorders) | 9 | 9 | 18
Eye pain - Study eye (Eye disorders) | 6 | 4 | 10
Eye pruritus - Fellow eye (Eye disorders) | 5 | 0 | 5
Eye pruritus - Study eye (Eye disorders) | 5 | 0 | 5
Macular fibrosis - Fellow eye (Eye disorders) | 2 | 4 | 6
Macular oedema - Fellow eye (Eye disorders) | 5 | 3 | 8
Vision blurred - Fellow eye (Eye disorders) | 0 | 4 | 4
Vision blurred - Study eye (Eye disorders) | 1 | 5 | 6
Visual acuity reduced - Fellow eye (Eye disorders) | 4 | 3 | 7
Visual acuity reduced - Study eye (Eye disorders) | 6 | 6 | 12
Vitreous floaters - Study eye (Eye disorders) | 4 | 4 | 8
Vitreous haemorrhage - Fellow eye (Eye disorders) | 5 | 6 | 11
Vitreous haemorrhage - Study eye (Eye disorders) | 2 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 10
Nausea (Gastrointestinal disorders) | 5 | 5 | 10
Vomiting (Gastrointestinal disorders) | 0 | 4 | 4
Asthenia (General disorders) | 3 | 7 | 10
Chest pain (General disorders) | 4 | 1 | 5
Oedema peripheral (General disorders) | 4 | 2 | 6
Peripheral swelling (General disorders) | 0 | 4 | 4
Pyrexia (General disorders) | 8 | 5 | 13
Bronchitis (Infections and infestations) | 7 | 5 | 12
COVID-19 (Infections and infestations) | 3 | 4 | 7
Conjunctivitis - Fellow eye (Infections and infestations) | 4 | 2 | 6
Conjunctivitis - Study eye (Infections and infestations) | 6 | 1 | 7
Gastroenteritis (Infections and infestations) | 4 | 0 | 4
Herpes zoster (Infections and infestations) | 2 | 5 | 7
Influenza (Infections and infestations) | 7 | 4 | 11
Nasopharyngitis (Infections and infestations) | 16 | 17 | 33
Pulpitis dental (Infections and infestations) | 2 | 4 | 6
Rhinitis (Infections and infestations) | 2 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 8
Urinary tract infection (Infections and infestations) | 5 | 4 | 9
Blood creatinine increased (Investigations) | 8 | 2 | 10
Blood pressure increased (Investigations) | 5 | 4 | 9
Blood triglycerides increased (Investigations) | 2 | 6 | 8
Blood urea increased (Investigations) | 3 | 4 | 7
Glycosylated haemoglobin increased (Investigations) | 7 | 5 | 12
Intraocular pressure increased - Fellow eye (Investigations) | 2 | 5 | 7
Intraocular pressure increased - Study eye (Investigations) | 6 | 4 | 10
Protein urine present (Investigations) | 4 | 5 | 9
White blood cells urine positive (Investigations) | 1 | 4 | 5
Gout (Metabolism and nutrition disorders) | 1 | 7 | 8
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 | 2 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Dizziness (Nervous system disorders) | 1 | 4 | 5
Headache (Nervous system disorders) | 8 | 4 | 12
Chronic kidney disease (Renal and urinary disorders) | 4 | 4 | 8
Diabetic nephropathy (Renal and urinary disorders) | 5 | 7 | 12
Proteinuria (Renal and urinary disorders) | 6 | 13 | 19
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 15
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 | 3 | 7
Hypertension (Vascular disorders) | 15 | 17 | 32
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03481660/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT03481660/SAP_001.pdf